CLINICAL TRIAL: NCT02167360
Title: A Phase II, Single Arm, Multicenter Trial to Determine the Efficacy and Safety of CTL019 in Adult Patients With Relapsed and Refractory B-cell Acute Lymphoblastic Leukemia
Brief Title: Study of Efficacy and Safety of CTL019 in Adult ALL Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not enroll
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: UPCC 07414
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-09

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Relapsed B-cell Acute Lymphoblastic Leukemia; Refractory B-cell Acute Lymphoblastic Leukemia
Keywords: adult patients; B-cell ALL; chemo-refractory; relapsed after allogeneic SCT; ineligible for allogeneic SCT
MeSH Terms: conditions — Burkitt Lymphoma | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: CTL019

INTERVENTIONS:
Drug: CTL019 — A dose of CTL019 transduced cells will consist of a single infusion of 2 to 10 x 108 CTL019 transduced cells.

SUMMARY:
This is a single arm, open-label, multi-center, phase II study to determine the efficacy and safety of CTL019 in adult patients with r/r B-cell ALL. The study will have the following sequential phases: Screening, Pre-Treatment, Treatment and Primary Follow-up, Secondary Follow-up (Relapse Follow-up) and Survival Follow-up. The total duration of the primary follow-up is 1 year from cell infusion. Safety will be assessed until the end of the treatment and primary follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory adult B-cell ALL a. First or greater Bone Marrow (BM) relapse OR b. Any BM relapse after allogeneic stem cell transplantation (SCT) and must be > 6 months from SCT at the time of CTL019 infusion OR c. Refractory as defined by not achieving a CR (morphology <5% blasts) after 2 cycles of a standard chemotherapy regimen OR d. Patients with Philadelphia chromosome positive (Ph+) ALL are eligible if they are intolerant to or have failed tyrosine kinase inhibitor therapy (TKI), or if TKI therapy is contraindicated.
* For relapsed patients, documentation of CD19 tumor expression in bone marrow or peripheral blood by flow cytometry within 3 months of screening
* Adequate organ function defined as:

  a. Renal function defined as: i. A serum creatinine of <1.5 x ULN OR ii. Calculated creatinine clearance or radioisotope Glomerular Filtration Rate (GFR) > 60 mL/min/1.73 m2 b. Alanine Aminotransferase (ALT) < 5 times the upper limit of normal (ULN) c. Bilirubin < 2.0 mg/dL d. Must have a minimum level of pulmonary reserve defined as ≤Grade 1 dyspnea and pulse oxygenation > 91% on room air e. Left Ventricular Ejection Fraction (LVEF) ≥ 45% confirmed by echocardiogram or Multiple Uptake Gated Acquisition (MUGA)
* Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening
* Age > 18 years
* A ECOG Performance Status that is either 0 or 1 at screening
* Signed written informed consent must be obtained prior to any study procedures
* Once all other eligibility criteria are confirmed, must have an apheresis product of non-mobilized cells received and accepted by the manufacturing site. Note: Apheresis product will not be assessed for acceptance by the manufacturing site until documented confirmation of all other eligibility criteria.
* Women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) must agree to use highly effective methods of contraception during the entire study period (1 year after the CTL019 infusion). Highly effective contraception methods include:

  1. Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are NOT acceptable methods of contraception)
  2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  3. Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient
  4. BOTH of the following forms of contraception must be utilized:

     * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
     * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  5. Use of intrauterine devices (IUD) are excluded due to increased risks of infection and bleeding in this population
  6. In case of use of oral contraception, women must be stable on the same pill for a minimum of 3 months before taking study treatment

Women who are not of reproductive potential (defined as post-menopausal for at least 24 consecutive months (i.e. have had no menses) or have undergone hysterectomy, salpingotomy, and/or bilateral oophorectomy) are eligible without requiring the use of contraception. Acceptable documentation includes written or oral documentation communicated by clinician or clinician's staff of one of the following:

1. Physician report/letter
2. Operative report or other source documentation in the patient record
3. Discharge summary
4. Follicle stimulating hormone measurement elevated into the menopausal range.

Exclusion Criteria:

* Isolated extra-medullary disease relapse
* Patients with concomitant genetic syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome.
* Patients with Burkitt's lymphoma/leukemia (i.e. patients with mature B-cell ALL, leukemia with B-cell [surface Immunoglobulin (sIg) positive and kappa or lambda restricted positivity] ALL, with French, American, British [FAB] L3 morphology and /or a MYC translocation)
* Prior malignancy, unless treated with curative intent and with no evidence of active disease present for > 5 years before screening
* Treatment with any prior gene therapy product
* Has had treatment with any prior anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy
* Active or latent hepatitis B or active hepatitis C, or any uncontrolled infection at screening 8. Human Immunodeficiency Virus (HIV) infection at screening 9. Presence of grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD) 10. The following medications are excluded:

  a. Steroids: Therapeutic doses of steroids must be stopped > 72 hours prior to CTL019 infusion. However, the following physiological replacement doses of steroids are allowed: < 6-12 mg/m2/day hydrocortisone or equivalent. Topical steroids are permitted.

  b. Allogeneic cellular therapy: Any donor lymphocyte infusions (DLI) must be completed > 6 weeks prior to CTL019 infusion c. GVHD therapies: Any drug used for GVHD must be stopped > 4 weeks prior to CTL019 infusion (e.g. calcineurin inhibitors, methotrexate or other chemotherapy drugs, mycophenolyate, University of Pennsylvania Page 20 of 138 Oncology Protocol Protocol No. UPCC#07414/CCTL019B2207J V00.1 04-02-2014 steroids [see above], rapamycin, thalidomide, or immunosuppressive antibodies such as rituximab, anti-tumor necrosis factor [anti-TNF] , anti-interleukin 6 [anti-IL6] or anti-interleukin 6 receptor [anti-IL6R]) d. Chemotherapy: i. The following drugs must be stopped >1 week prior to CTL019 infusion: hydroxyurea, vincristine, 6-mercaptopurine, 6-thioguanine, methotrexate <25 mg/m2, cytosine arabinoside <10 mg/m2/day, asparaginase ii. The following drugs must be stopped >4 weeks prior to CTL019 infusion: salvage chemotherapy (e.g. clofarabine, cytosine arabinoside >100mg/m2, anthracyclines, cyclophosphamide), excluding the required lymphodepleting chemotherapy drugs e. CNS disease prophylaxis i. CNS prophylaxis treatment must be stopped > 1 week prior to CTL019 infusion (e.g. intrathecal methotrexate).

  11. Active Central Nervous System (CNS) involvement by malignancy, defined as CNS-3 per National Comprehensive Cancer Network (NCCN) guidelines. Note: Patients with history of CNS disease that has been effectively treated will be eligible.

  12. Patient has received an investigational medicinal product within the last 30 days prior to screening 13. Pregnant or nursing (lactating) women. NOTE: female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01-11 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Frey, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine